CLINICAL TRIAL: NCT04360239
Title: Stopping Fish Oil Supplementation Prior to Total Hip Replacement a Randomized Clinical Trial
Brief Title: Fish Oil in Total Hip Replacement Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey L Stimac MD (Other)
Responsible Party: Sponsor-Investigator, Jeffrey L Stimac MD, Principal Investigator, Norton Healthcare
Organization: Norton Healthcare (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-N0364
Record Dates: First submitted 2020-03-05; First posted 2020-04-24 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2022-06

CONDITIONS: Total Hip Arthroplasty
Keywords: Fish Oil; Total Hip Arthroplasty; Blood management; Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fish Oil (Experimental): Fish-Oil naïve subjects will be started on fish oil 4 weeks prior to surgery and continued until the 6 week follow up. Subjects already taking fish oil will be switched to the study fish-oil formulation of two capsules twice daily (3000 mg of EPA and DHA).
  Interventions: Dietary Supplement: Fish Oil
- Control (No Intervention): No fish oil supplementation

INTERVENTIONS:
Dietary Supplement: Fish Oil — Fish-oil formulation of two capsules twice daily (3000 mg of EPA and DHA).
  Arms: Fish Oil

SUMMARY:
The purpose of this study is to determine if continuing fish oil supplementation leads to higher blood loss in patients undergoing total hip arthroplasty (THA). Another purpose is to determine if patients on fish oil have less pain after THA. Fish oil (Omega-3 fatty acid) is commonly used by patients as a natural anti-inflammatory to decrease joint pain from arthritis. Supplements, including fish oil, are typically stopped 1-2 weeks prior to surgery as there is an increased risk of perioperative bleeding. However, there are current methods in joint replacement surgery that decrease the risk of perioperative bleeding. With the risk of excessive bleeding being minimized, fish oil may not need to be stopped prior to surgery and could be continued immediately after surgery. The anti-inflammatory effect of fish oil may also help decrease pain after surgery.

DETAILED DESCRIPTION:
Introduction/Purpose Fish oil (Omega-3 fatty acid) is commonly used by patients as a natural anti-inflammatory to decrease joint pain from arthritis. Furthermore, fish oil has been found to decrease the risk of coronary artery disease, decrease mild hypertension, prevent cardiac arrhythmias and decrease blood triglyceride levels. Supplements, including fish oil, are typically stopped 1-2 weeks prior to surgery as there is an increased risk of perioperative bleeding. With modern blood management techniques in joint replacement surgery, including the use of tranexamic acid, the risk of perioperative bleeding may be minimized. With the risk being minimized fish oil may not need to be stopped prior to surgery and could be continued immediately after surgery. The anti-inflammatory effect of fish oil in the perioperative period may aid in post-operative pain management. The purpose of this study is to determine if continuing fish oil supplementation leads to higher blood loss in patients undergoing unilateral total hip arthroplasty (THA). A secondary analysis is to determine if patients on fish oil have less pain after THA.

Objectives

Primary Outcome Measures:

• Calculated total perioperative blood loss milliliters (mL) using Bourke's, Gross', Camarasa's, and Lopez-Picado's formula based on post-operative (PO) D5 Hemoglobin and Hematocrit

Secondary Outcomes Measures:

* Incidence of blood transfusion
* Post-operative day 1 Hemoglobin and Hematocrit
* Post-operative pain scores
* Pain medication usage (morphine equivalents)
* Difference in wound complications (superficial and deep infection, drainage, hematoma)

Study Design Open-label, adaptive randomized clinical trial with a 1:1 randomization

Study arms:

Control: No fish oil supplementation. Interventional: Fish oil supplementation started or continued Fish-Oil naïve subjects will be started on fish oil 4 weeks prior to surgery and continued until the 6 week follow up. Subjects already taking fish oil will be switched to the study fish-oil formulation of two capsules twice daily (3000 mg of EPA and DHA).

All subjects will be asked to stop all non-Fish Oil supplements 2 weeks prior to and 2 weeks after surgery.

Sample size: The primary outcome is blood loss, mean of 1200 mL with a reported standard deviation of 340 mL. A non-inferiority trial to determine if there is no difference in blood loss between subjects taking fish oil and subjects not taking fish-oil will require 50 subjects in each arm with 80% power lower limit of a one-sided 90% confidence two-sided confidence interval that the difference between the two groups is one half the reported standard deviation of 340 mL (170 mL). To allow for drop-outs, 60 subjects will be enrolled in each arm.

Randomization: As patients already taking fish-oil supplements will likely not be willing to discontinue their regimen, an adaptive randomization will be performed. Patients already on fish-oil will be assigned to the Interventional Arm and the subsequent randomization adjusted.

Study Procedures After being deemed eligible, potential study participants will be approached about the study asked to sign an informed consent form that has been approved by the internal review board. Patients that meet the inclusion criteria will be randomized to either the control group or experimental group. Patients in the experimental group will started on 3000 mg of EPA and DHA 4 weeks prior to surgery. The fish oil will be continued in the perioperative period and until their 6 week follow up appointment. Patients will be supplied the fish oil at no cost. Patients will stop all other supplements and herbal medicines 2 weeks prior to surgery and will not restart the supplements until 2 weeks after surgery.

Pre-operative hemoglobin and hematocrit will be obtained on all patients during preadmission testing. All patients must stay one night in the hospital after surgery. A post-day #1 and #5 hemoglobin and hematocrit will be obtained on all patients. Amount of fluid collected in the wound drain will also be collected. Blood loss will be calculated using the Bourke's, Gross', Camarasa's, and Lopez-Picado's formula. Data will be collected on the rates of blood transfusions for each patient. Post-operative day 1 pain scores will be determined for each patient using the visual analog scale. Pain medication use through patient report will be collected and daily morphine equivalents starting on the day of surgery up until the patients 6 week follow up will be calculated. Date and quantity of any narcotic refill will be recorded. Data will also be collected on the rate of wound complications in patients. Enrollment into the study is voluntary and participants can voluntarily withdraw at any time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Primary total hip arthroplasty
* Diagnosis of osteoarthritis
* Able to consume fish oil
* Medically cleared for surgery
* Plan for unilateral total hip arthroplasty
* Able to consent to surgery and study participation

Exclusion Criteria:

* Unable to consent for study participation
* Unable to participate in preoperative testing
* History of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* Patient reports of easy bruising
* Revision total hip replacement
* Indication for surgery other than osteoarthritis
* History of surgical wound complication on involved extremity
* Allergy to fish oil
* Allergy to Aspirin
* Patients on Coumadin, Eliquis, Xarelto or other anticoagulants (excluding NSAIDs)
* Outpatient total hip replacement
* Bilateral total hip replacement
* Coagulopathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Total perioperative blood loss | Post-operative day 5
  Calculated total perioperative blood loss (mL) using Bourke's, Gross', Camarasa's, and Lopez-Picado's formula based on Post Operative Day 5 (POD5) Hemoglobin and Hematocrit

SECONDARY OUTCOMES:
Post-operative day 1 Hemoglobin | Post-operative day 1
  Post-operative day 1 Hemoglobin
Post-operative day 1 Hematocrit | Post-operative day 1
  Post-operative day 1 Hematocrit

OTHER OUTCOMES:
Post-operative pain scores | Post-operative day 1 pain scores will be determined for each patient using the visual analog scale
  Post-operative pain scores will be determined for each patient using a numeric rating scales (NRS) with 0 being no pain and 10 being worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Stimac, MD, Principal Investigator — Norton Healthcare
Locations (1):
- Norton Healthcare, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akintoye E, Sethi P, Harris WS, Thompson PA, Marchioli R, Tavazzi L, Latini R, Pretorius M, Brown NJ, Libby P, Mozaffarian D. Fish Oil and Perioperative Bleeding. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e004584. doi: 10.1161/CIRCOUTCOMES.118.004584. PMID 30571332
- [Background] Boe C, Vangsness CT. Fish Oil and Osteoarthritis: Current Evidence. Am J Orthop (Belle Mead NJ). 2015 Jul;44(7):302-5. PMID 26161757
- [Background] Calder PC. Omega-3 fatty acids and inflammatory processes: from molecules to man. Biochem Soc Trans. 2017 Oct 15;45(5):1105-1115. doi: 10.1042/BST20160474. Epub 2017 Sep 12. PMID 28900017
- [Background] Connor SL, Connor WE. Are fish oils beneficial in the prevention and treatment of coronary artery disease? Am J Clin Nutr. 1997 Oct;66(4 Suppl):1020S-1031S. doi: 10.1093/ajcn/66.4.1020S. PMID 9322583
- [Background] Kremer JM. Fish Oil and Inflammation - A Fresh Look. J Rheumatol. 2017 Jun;44(6):713-716. doi: 10.3899/jrheum.161551. No abstract available. PMID 28572471
- [Background] Tummala R, Ghosh RK, Jain V, Devanabanda AR, Bandyopadhyay D, Deedwania P, Aronow WS. Fish Oil and Cardiometabolic Diseases: Recent Updates and Controversies. Am J Med. 2019 Oct;132(10):1153-1159. doi: 10.1016/j.amjmed.2019.04.027. Epub 2019 May 8. PMID 31077653